CLINICAL TRIAL: NCT03521843
Title: Study of Local Drug Delivery in the Treatment of Femoropopliteal In-stent Restenosis
Brief Title: LDD in Treatment of Femoropopliteal ISR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12345678
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Peripheral Artery Disease; In-stent Restenosis
Keywords: femoropopliteal occlusive disease; local drug delivery; endovascular treatment
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: only the doctors know the group the patient goes into
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- balloon dilation only (Experimental): The balloon dilation only will be used to treat the femoropopliteal in-stent restenosis.
  Interventions: Device: balloon dilation only
- balloon dilation+local drug delivery (Experimental): The balloon dilation and local drug delivery will be used to treat the femoropopliteal in-stent restenosis.
  Interventions: Device: balloon dilation+local drug delivery

INTERVENTIONS:
Device: balloon dilation only — The balloon dilation only will be used to treat the femoropopliteal in-stent restenosis.
  Arms: balloon dilation only
Device: balloon dilation+local drug delivery — The balloon dilation and local drug delivery will be used to treat the femoropopliteal in-stent restenosis.
  Arms: balloon dilation+local drug delivery

SUMMARY:
This study will evaluate the effectiveness and safety of local drug delivery using TAPAS balloon catheter system in the treatment of femoropopliteal in-stent restenosis. Patients with femoropopliteal in-stent restenosis will randomly receive balloon dilation or balloon dilation plus local drug delivery using balloon catheter system. Their clinical outcomes (e.g. 12-month late lumen loss or late lumen loss at secondary intervention within 12 months, 6-month and 1-year patency rate of target vessel) in 1 year after the treatment will be compared.

DETAILED DESCRIPTION:
Femoropopliteal occlusive disease is a common type of peripheral arterial disease. Endovascular treatment has been the first-line treatment of femoropopliteal occlusive disease. However, the in-stent re-stenosis has been a major limitation of well long-term patency after stent implantation. The chronic inflammation induced by stenting could be a main reason of restenosis. Then the concept "leave nothing behind" is proposed, and some novel treatment methods and devices are developed. Here, the investigators propose the hypothesis that using local drug delivery with TAPAS balloon system can relieve the inflammation induced by the stent implantation and balloon dilation. Therefore, 40 patients of femoropopliteal in-stent restenosis will be randomly allocated into the group "balloon dilation+local drug delivery with balloon system" or "balloon dilation only". The 1-year patency rate,12-month late lumen loss, incidence of complications, imaging parameters will be compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* have signed the informed consent
* age of 18-80 years old
* femoropopliteal artery disease (Rutherford 2-4)
* femoropopliteal in-stent restenosis (≥70%)
* length of lesion ≤ 20cm
* at least one infrapopliteal run-off vessel

Exclusion Criteria:

* serum Cr > 150 umol/L
* patients with acute thrombosis
* stent fracture within femoropopliteal artery
* allergic to aspirin, heparin, clopidogrel, paclitaxel, contrast medium
* already recruited into other clinical trials that could influence the outcome of this study
* pregnancy and lactation
* relatively easy bleeding
* malignancy or irreversible organ failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
target lesion revascularization | 12 months
  the revascularization rate of target lesion

SECONDARY OUTCOMES:
MLD | 6 months
  minimal lumen diameter of target vessel at 6 months
restenosis rate | 6 months
  the rate of re-stenosis (≥50) of target vessel at 6 months
adverse events | 12 months
  incidence of treatment related adverse events
Rutherford level | 12 months
  change of Rutherford level
ABI | 12 months
  change of ankle brachial index
main amputation | 12 months
  rate of main amputation
12-month patency rate | 12 months
  the 12-month patency rate of target vessel
6-month patency rate | 6 months
  the 6-month patency rate of target vessel
late lumen loss rate at secondary intervention | 12 months
  the rate of late lumen loss of target vessel at secondary intervention within 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China